CLINICAL TRIAL: NCT02699853
Title: Prospective Randomized Comparison of Robotic Versus Open Radical Cystectomy
Brief Title: Robotic or Open Radical Cystectomy in Treating Patients With Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to revamp the protocol completely and will submit as new study.
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4B-15-4; NCI-2016-00080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-15-00731; 4B-15-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Stage 0is Bladder Urothelial Carcinoma; Stage I Bladder Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma; Stage III Bladder Urothelial Carcinoma
MeSH Terms: interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (RRC) (Experimental): Patients undergo RRC at day 0.
  Interventions: Other: Questionnaire Administration; Procedure: Radical Cystectomy
- Arm II (ORC) (Experimental): Patients undergo ORC at day 0.
  Interventions: Other: Questionnaire Administration; Procedure: Radical Cystectomy

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Radical Cystectomy — Undergo RRC
  Other Names: Complete Cystectomy
  Arms: Arm I (RRC)
Procedure: Radical Cystectomy — Undergo ORC
  Other Names: Complete Cystectomy
  Arms: Arm II (ORC)

SUMMARY:
This randomized phase II trial studies how well robotic radical cystectomy (RRC) or open radical cystectomy (ORC) works in treating patients with bladder cancer. Cystectomy is a surgical procedure to remove all or part of the bladder (the organ that holds urine) or to remove a cyst (a sac or capsule in the body). In RRC, the the surgeon makes small cuts in the abdomen and uses a thin, lighted instrument with a camera attached called a scope. With the help of a robot, the surgeon removes the bladder and other nearby structures. In ORC, the surgeon makes a cut into the lower abdomen to expose the urinary tract in order to remove the bladder and nearby structures. It is not yet known whether RRC or ORC has fewer complications, better quality of life, and faster recovery time in treating patients with bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare RRC to ORC in terms of the difference in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core (QLQC)30 quality of life instrument assessed at baseline to day 30 after radical cystectomy (RC).

II. To compare RRC to ORC in terms of the 90-day high-grade complication rate (where high grade is defined as Clavien-Dindo grade 3-5).

III. To compare the peri-operative cost of the RC procedure, as defined as from the day of hospital admission to the day of hospital discharge.

SECONDARY OBJECTIVES:

I. To estimate the differences between RRC and ORC in terms of the following quality of life outcomes: Narcotic requirements prior to RC, during hospital stay and on days 7, 14, 30, 6 weeks, and 3, 6, 9 and 12 months; Visual Analog Scale (VAS) pain score prior to RC and on days 7, 14, 30, 6 weeks, and 3, 6, 9 and 12 months; the EORTC-QLQ-30 prior to RC and at 3, 6, 9, and 12 months; the bladder cancer index (BCI) at 30 days and 3, 6, 9, and 12 months; the Sexual Health Inventory for Men (SHIM) prior to RC and at 3, 6, 9, and 12 months; the World Health Organization (WHO) Quality of Life (QOL) questionnaire prior to RC and at 30 days and 3, 6, 9, and 12 months.

II. To estimate the differences between RRC and ORC in terms of the following surgical and complication outcomes: all complications occurring intraoperatively, during postoperative hospitalization and during the 90 days post cystectomy assessed at 7, 14, and 30 days; at 6 weeks and at 3 months-graded according to the Clavien-Dindo classification; all complications, all grade 3+ complications, and all grade 4+ complications; time to oral intake; estimated blood loss during surgery, number of transfusions on the day of surgery; drop in hematocrit at 24 hours; lymph node yield; and positive surgical margin.

III. To estimate the differences between RRC and ORC in terms of the following cost-related outcomes: operation room time; number of disposables used; pharmacy costs; length of hospital stay; admission to intensive care unit (ICU) prior to discharge & length of stay in ICU; number of hospital readmissions within 30 and 90 days (3 months); necessary tests/procedures to treat complications during hospitalization and within 30 and 90 days.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo RRC at day 0.

ARM II: Patients undergo ORC at day 0.

After completion of study treatment, patients are followed up at 7 days, 30 days, 6 weeks, and at 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radical cystectomy for urothelial cancer
* All types of urinary diversions
* Tis-T3 Urothelial cancer; patients will be stratified according to clinical stage
* Ability to consent
* Patient meets criteria to be a surgical candidate

Exclusion Criteria:

* Inability to give consent or adhere to follow-up schedule
* T4 tumor
* Bulky lymphadenopathy (> 2 cm)
* Prior pelvic radiation
* Not surgical candidate because of significant co-morbidity
* Uncontrolled coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Change in patient reported quality of life, as measured by the EORTC-QLQ-C30 | Baseline and 1-month post cystectomy
  The results for the two arms will be summarized using graphical methods and standard descriptive statistics. Means (or medians) and associated 95% confidence intervals-for each arm separately and for the difference-will be used to display the patterns. For QoL variables that are assessed at multiple times post cystectomy, regression methods that accommodate repeated measures will be used to assess patterns over time. Analyses will compare the two arms using general linear regression models and stratifying for the four variables used for stratification prior to randomization.

SECONDARY OUTCOMES:
Change in erectile dysfunction, as measured by the SHIM score | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Desai, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States